CLINICAL TRIAL: NCT06104579
Title: Quality Check: Concordance Between Two Monitoring Systems for Postoperative Organ/Space Surgical Site Infections in Rectal Cancer Surgery. Linkage of Data From the Catalan Cancer Plan (CCP) and the Catalan Healthcare-associated Infections Surveillance Programme (VINCat).
Brief Title: Concordance Between Monitoring Systems for Organ/Space Surgical Site Infections in Rectal Surgery
Status: Completed | Type: Observational
Sponsor: Hospital de Granollers (Other)
Collaborators: Institut d'Investigació Biomèdica de Bellvitge (Other); Institut Català d'Oncologia (Other)
Responsible Party: Sponsor
Other Study IDs: VINCat_PDO
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2023-10

CONDITIONS: Rectal Cancer; Organ-Space Surgical Site Infection
Keywords: Surgical Site Infection; Rectal cancer; Rectal Surgery; Databases concordance
MeSH Terms: conditions — Rectal Neoplasms; Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients operated on rectal cancer, included in the Catalan Cancer Registry: Patients operated on rectal cancer, included in two compulsory audits of the Catalan Cancer registry, and who suffered an organ-space surgical infection.
  Interventions: Other: Person-level linkage of both databases looking for concordance in the diagnosis of organ-space surgical site infection
- Patients operated on rectal surgery, included in the Catalan Infection Surveillance Program: Patients included in the voluntary Catalan Infection Surveillance Program, and followed for 30 days postoperatively, and who suffered an organ-space surgical infection.
  Interventions: Other: Person-level linkage of both databases looking for concordance in the diagnosis of organ-space surgical site infection

INTERVENTIONS:
Other: Person-level linkage of both databases looking for concordance in the diagnosis of organ-space surgical site infection — Concordance between the two registers was analysed using Cohen´s Kappa.

SUMMARY:
The Catalan Cancer Plan (CCP) undertakes periodic audits of cancer treatment outcomes, including organ/space surgical site infections (O/S-SSI) rates, while the Catalan Healthcare-associated Infections Surveillance Programme (VINCat) carries out standardized prospective surveillance of surgical site infections (SSIs) in colorectal surgery. This cohort study aimed to assess the concordance between these two monitoring systems for O/S-SSI following primary rectal cancer surgery.

DETAILED DESCRIPTION:
The healthcare system in Catalonia (Spain) monitors and reports SSI in cancer patients through two principal mechanisms. First of all, the Catalan Cancer Plan (CCP) is a Health Department structure that aims to improve the quality of care for cancer patients by means of periodic auditing of outcomes with real-world data and feedback to professionals. One indicator included in these compulsory audits is the occurrence of O/S-SSI.

On the other hand, the Catalan Healthcare-associated Infections Surveillance Programme (VINCat) is a nationwide network for hospital-acquired infections (HAI) which conducts surveillance in colorectal surgery.

The two systems thus operate with an important difference: the CCP audits are mandatory and cover all cancer surgeries performed in centres funded through the public healthcare system, while VINCat is a voluntary registry programme among participating centres. The selected cases and methods used to detect O/S-SSI may therefore vary substantially between auditing systems.

This retrospective population-based cohort study aims to assess the concordance between clinical audits of the CCP and the VINCat registry as a preliminary step to studies correlating local recurrence after rectal cancer surgery and O/S-SSI.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old
* Eligible patients with tumour ≤ 13 cm from anal verge, as measured by Magnetic Resonance Imaging
* Primary adenocarcinoma
* Oncological resection with curative intent
* Cancer stages: I-II-III

Exclusion Criteria:

* Transanal local resection
* Emergency colorectal surgeries
* Presence of metastases found in the diagnostic process or during the surgical procedure
* Recurrence of the disease treated before the study period
* Non-resectable tumour or palliative surgery
* Patients operated in private centres

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated on rectal surgery for rectal cancer in Catalonia, Spain.
Sampling Method: Non-Probability Sample
Enrollment: 11367 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Rate of Organ-space surgical site infection | 30 days
  As described by the Centers for Disease Control: an infection occurring within 30 days of the surgical procedure and involves any part of the body deeper than the fascial/muscle layers that is opened or manipulated during surgery. In addition, the patient must present at least one of the following associated events: a purulent drainage from a drain placed into the organ/space

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Català d'Oncologia, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
: Restrictions apply to the availability of these data, which belong to two national databases and are not publicly available. Data was obtained from the Catalan Cancer Plan and VINCat, and are only available with the permission of their Technical Committees.

REFERENCES:
- [Derived] Matallana C, Pera M, Espin-Basany E, Biondo S, Badia JM, Limon E, Pujol M, de Lacy B, Aliste L, Borras JM, Manchon-Walsh P. Quality check: concordance between two monitoring systems for postoperative organ/space-surgical site infections in rectal cancer surgery. Linkage of data from the Catalan Cancer Plan and the VINCat infection surveillance programme. World J Surg Oncol. 2024 May 25;22(1):138. doi: 10.1186/s12957-024-03410-9. PMID 38789966